CLINICAL TRIAL: NCT04114838
Title: Cohort Study of Patients Treated for Peripheral Arterial Occlusive Disease
Acronym: EndoRevI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EndoRevI
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Obstructive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral Arterial Occlusive Disease is associated with a high risk of cardiovascular events. The critical ischemia stage represents the most severe stage of Peripheral Arterial Occlusive Disease, associated with decubitus pain and / or foot ulceration. The severity of this arterial involvement involves functional prognosis of the lower limb with a high risk of amputation, and the vital prognosis of the patient. In these patients, the rate of amputation and mortality at 1 year can reach 20%. Therefore, the goal of management in a multidisciplinary setting is limb salvage and improvement of the patient's vital prognosis.

In the vascular medicine department, the indication and modalities of the revascularization procedure are discussed in a multidisciplinary consultation meeting. Surgical revascularization by distal bypass requires venous material that can be used, a receiving artery without diffuse lesions, in direct continuity with the arterial network of the foot, and the absence of co-morbidities against general anesthesia. With the modernization and development of endovascular equipment dedicated to the hamstrings, the interventional radiology techniques in the management of critical ischemia allow the treatment of one or more arterial axes as well as a very distal revascularization in the arteries. of the foot with less morbidity-mortality compared to surgery, especially in patients the most fragile patients. Since 2013, the endovascular revascularization procedures performed by the interventional radiology team have been an integral part of the management of patients with peripheral arterial disease of the lower limbs monitored in the vascular medicine department. The hospital is therefore a privileged place to observe the long-term impact of this medical care on the future of patients with different stages of severity of arterial disease.

The objective of this retrospective study is to evaluate the life-threatening, limb salvage and associated prognostic factors in patients with Peripheral Arterial Occlusive Disease supported by endovascular revascularization in the vascular medicine department of the GHPSJ.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with intermittent / intermittent claudication / arterial ulcer / mixed ulcer / critical ischemia / acute ischemia, whose need for a revascularization procedure in the patient's medical management was discussed and confirmed as a multidisciplinary staff between 1st November 2013 and September 2018
* endovascular revascularized Patient
* Francophone patients

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients who oppose the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were hospitalized the vascular medicine department of the Hospital Group Paris Saint-Joseph, for management of an PAOD with endovascular revascularization, between November 1, 2013 and September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Survival rate without major amputation | year 1
  The outcome measure the survival rate without major amputation at 1 year.

SECONDARY OUTCOMES:
Prevalence of Intraoperative Deaths and Cardiovascular Events | Day 1
  This measures the prevalence of Intraoperative Deaths and Cardiovascular Events.
Prevalence of Deaths and Cardiovascular Events, at 1 month | Month 1
  This measures the prevalence of Deaths and Cardiovascular Events, 1 month after the surgery.
Prevalence of Deaths and Cardiovascular Events, at 1 year | Year 1
  This measures the prevalence of Deaths and Cardiovascular Events, 1 year after the surgery.
Healing rate | Year 1
  This outcome measure the healing rate, 1 year after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra YANNOUTSOS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Yannoutsos A, Lin F, Billuart O, Gaisset R, Sacco E, Beaussier H, Buronfosse A, Mourad JJ, Emmerich J, Lazareth I, Priollet P. Predictive value of admission blood pressure for 3-month mortality in patients undergoing revascularization for critical limb ischemia. J Hypertens. 2020 Dec;38(12):2409-2415. doi: 10.1097/HJH.0000000000002556. PMID 32694333